CLINICAL TRIAL: NCT00945932
Title: A Randomised, Double-blind, Placebo-controlled, 2-way Crossover Study to Determine the Efficacy of Repeat Inhaled Doses of GW870086X on FEV1 in Mild to Moderate Asthmatics
Brief Title: A Study to Evaluate the Effect of Repeat Doses of GW870086X in Mild to Moderate Asthmatics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 112851
Record Dates: First submitted 2009-07-16; First posted 2009-07-24 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: asthma; GW870086X; Efficacy; FEV1; repeat-dose
MeSH Terms: conditions — Asthma | interventions — GW870086X

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 28 day repeat dose (Experimental)
  Interventions: Drug: GW870086X; Drug: Placebo

INTERVENTIONS:
Drug: GW870086X — Investigational product
Drug: Placebo — Placebo control

SUMMARY:
This study will measure the effect of repeat inhaled doses of GW870086X on lung function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and oestradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 90-95 hours post-last dose.
* Body weight, men >/= 50 kg, women >/= 45 kg and BMI within the range 19.0 - 29.0 kg/m2 (inclusive).
* Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit and currently being treated only with intermittent short-acting beta-2 agonist therapy by inhalation.
* Severity of Disease: A best FEV1 of 40%-85% of the predicted normal value during the Visit 1 screening period.
* No history of smoking within 6 months of the start of the study, and with a total pack year history of </= 10 pack years
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin </= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* Subject is mentally or legally incapacitated.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, bronchiectasis or pulmonary fibrosis).
* Clinically significant abnormalities in safety laboratory analysis at screening.
* Subject has known history of hypertension or is hypertensive at screening. Hypertension at screening is defined as persistent systolic BP >140mmHg or diastolic BP > 90mmHg.
* Respiratory tract infection and/or exacerbation of asthma within 4 weeks prior to the first dose of study medication.
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest and/or hypoxic seizures.
* Administration of oral, injectable or dermal steroids within 8 weeks of screening.
* Administration of intranasal and/or inhaled steroids within 2 week of the screening visit. Prior to this the subject's maximum daily dose must be less than FP equivalent 250mcg.
* Respiratory Infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within the 4 weeks before screening and led to a change in asthma management, or in the opinion of the Investigator is expected to affect the subjects asthma status or the subjects ability to participate in the study.
* Asthma Exacerbation: Any asthma exacerbation requiring oral corticosteroids within 8 weeks of screening. A subject must not have had any hospitalisation for asthma within 6 months prior to screening
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Paracetamol is an exception and will be permitted at daily doses of up to 4 g from screening to follow-up.
* Has taken Xanthines (including theophylline, but not including caffeine), anticholinergics, cromoglycates and/or long-acting beta-2 agonists within 1 week prior to screening and is unable to abstain from them throughout the study.
* Unable to abstain from other medications including non-steroidal anti-inflammatory drugs (NSAIDs), anti-depressant drugs, anti-histamines and anti-asthma (not including steroids), anti-rhinitis or hay fever medication, other than short acting inhaled beta-2 agonists and paracetamol (up to 4 g per day) for the treatment of minor ailments eg headache from 7 days before screening until the follow-up visit.
* Unable to abstain from medication or supplements that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, including ritonavir and ketoconazole from screening and throughout the study.
* Unable to use the DISKHALER device correctly.
* History of sensitivity to any of the study medications (including lactose), or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 ml within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects who are kept due to regulatory or juridical order in an institution.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Lung function as measured by FEV1 | Day 28

SECONDARY OUTCOMES:
Lung function as measured by FEV1 | Day 7 and 14
Lung function as measured by PEFR | Twice daily over 28 days
Rescue medication usage | 4-5 months
Assess safety and tolerability | 4-5 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (5):
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bareille P, Hardes K, Donald AC. Efficacy and safety of once-daily GW870086 a novel selective glucocorticoid in mild-moderate asthmatics: a randomised, two-way crossover, controlled clinical trial. J Asthma. 2013 Dec;50(10):1077-82. doi: 10.3109/02770903.2013.837480. Epub 2013 Oct 1. PMID 23991670
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 112851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112851 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register